CLINICAL TRIAL: NCT05643846
Title: Quadratus Lumborum Block After Cesarean Section: Analgesic Efficacy of Different Concentrations of Local Anesthetics. A Randomized Clinical Trial
Brief Title: Quadratus Lumborum Block After Cesarean Section: Analgesic Efficacy of Different Concentrations of Local Anesthetics
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danat Al Emarat Hospital (Other)
Responsible Party: Principal Investigator, JINAN AHMED JAMEEL AL ALOOSI, Principle Investigator, Danat Al Emarat Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RP DAE/2022/102
Record Dates: First submitted 2022-10-27; First posted 2022-12-09 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Outcome Measures

STUDY DESIGN:
Intervention Model Description: It is a Prospective, Double-blinded, randomized and controlled clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants are allocated randomly by means of computer generation sequencing. The allocation sequence with unique study number for each participant will be concealed in sequentially numbered, opaque, sealed, and stapled envelopes. This envelope will be opened by an anesthetist who was not involved in the study. This Anesthetist prepares the study medication as per the allocation and labels the syringe with the unique study number; this number will be used to identify the study medication and will be revealed only on completion of data collection at the end of the study. The investigators, participants and other healthcare providers who are involved in postoperative care, are blinded to the participant's group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Group 1) will receive the intervention 'Bupivacaine at concentration of 0.125%, dose of 0.2 ml/kg'. (Active Comparator): (Group 1) will receive bilateral QLB procedure with the intervention 'Bupivacaine local anesthetic drug at concentration of 0.125% concentration, at a dose of 0.2 ml/kg'.
  Interventions: Procedure: QLB procedure after cesarean section
- (Group 2) will receive the intervention 'Bupivacaine concentration of 0.25%, dose of 0.2 ml/kg'. (Active Comparator): (Group 2) will receive bilateral QLB procedure with the intervention 'Bupivacaine local anesthetic drug at a concentration of 0.25% concentration, at a dose of 0.2 ml/kg'.
  Interventions: Procedure: QLB procedure after cesarean section

INTERVENTIONS:
Procedure: QLB procedure after cesarean section — Bupivacaine local anesthetic drug used for QLB procedure after Cesarean section. Intervention of two different concentration of Bupivacaine, 0.125% or 0.25%, at a dose of 0.2 ml/kg.
  Other Names: Bupivacaine Local anesthetic drug at concentrations of 0.125% or 0.25%; Marcaine local anesthetic drug at concentration of 0.125% or 0.25%, at a dose of 0.2ml/kg

SUMMARY:
QLB is an injection of a local anesthetics around the quadratus lumborum muscle. It uses a fascial compartment path to extend the distribution of local anesthetics into the posterior abdominal wall and paravertebral space. This central effect can be of vital importance when managing the visceral pain after caesarean section.

Many studies have shown that the inclusion of quadratus lumborum block to a multimodal analgesic regimen would reduce pain scores, opioid consumption, and prolonging time to first rescue analgesic after cesarean delivery.

However, the dose and concentration of the local anesthetic used among the studies are varied, and literature search identified no randomized controlled trial which looked at the concentration -response of local anesthetic to optimize the concentration resulting in the best pain relief.

It is a perspective randomized controlled trial to compare the analgesic efficacy of 2 different concentrations of Bupivacaine to standardize postoperative analgesic protocol used for QLB after caesarean section.

DETAILED DESCRIPTION:
QLB is an injection of a local anesthetics around the quadratus lumborum muscle. It uses a fascial compartment path to extend the distribution of local anesthetics into the posterior abdominal wall and paravertebral space. Acute post C-section pain is a leading anesthetic concern for women; a key determinant of maternal satisfaction; may lead to persistent postoperative pain; is a predictor of postpartum depression; and can reduce early breastfeeding success. Effective postoperative analgesia should, therefore, be prioritized to improve outcomes following caesarean delivery. This study is a Double-blinded, randomized and controlled trial.

A written, informed consent is discussed with and signed by all participants, and the participants are randomly assigned into one of two groups; (Group 1) to receive bilateral QLB with '0.125% bupivacaine 0.2 ml/ kg', (Group 2) to receive bilateral QLB with '0.25% bupivacaine 0.2 ml/kg'. For all participants, spinal anesthesia is performed with ultrasonography guidance in a standardized manner using hyperbaric bupivacaine 15mg and fentanyl 25 μg.

At the end of the procedure in the supine position, all participants receive bilateral QLBs performs under ultrasound guidance and aseptic technique. The internal oblique muscle is identified and followed laterally to the lateral interfacial triangle sitting above the quadratus lumborum muscle.

Results will be reported as

1. Total number of PCA morphine demands and the actual doses delivered at predetermined time intervals (1h, 2 h, 4h, 6 h, 12 h, 24 h and 48 h) after surgery
2. Record of supplemental and regular analgesics.
3. Visual analogue score for pain at rest (static) and with movement (dynamic) (defined as the elevation of the head and shoulders off the pillow from the supine position), (0, no pain; 10, worst pain imaginable).
4. Residual nerve block (the time to mobilization)
5. Block-related complications (i.e., hematoma, organ injury, local anesthetic systemic toxicity, and sepsis).

6- Opioids-related side effects (Nausea, Vomiting, Itching)

The investigators hypothesized that using a higher concentration (0.25%) of local anesthetic (Bupivacaine) would increase the analgesic effect without increasing the side effects and complications.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are American Society of Anesthesiologists physical status 1 or 2.
* Participants who have singleton pregnancy at a gestation of at least 37 weeks.
* Participant who are scheduled for elective caesarean section under spinal anesthesia.
* Participants who are consented to be enrolled into the study.

Exclusion Criteria:

* Patients who have contraindications to spinal or regional anesthesia (Coagulopathy or on anticoagulants).
* Who have Allergy or sensitivity to study medications.
* Who have anatomical abnormalities or localized infection.
* Who have history of chronic pain or on regular opioids use.
* Who are unable to comprehend or unable to use the verbal rating pain scoring system,
* Failed spinal anesthesia or conversion to general anesthesia after spinal anesthesia.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 196 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2025-09-06 (Estimated); Study Completion 2025-12-06 (Estimated)

PRIMARY OUTCOMES:
Morphine dose requirements for pain control after surgery | Day 0, Day1, Day 2 after surgery.
  Actual doses of PCA morphine, in milligram unit, delivered to the participant after surgery on Day 0, Day1, and on Day2 after surgery.
Total number of morphine demands after surgery. | Day 0, Day1, Day 2 after surgery.
  Total number of PCA morphine demands after surgery on Day 0, on Day1, and on Day2 after surgery.
Assessment of heart rate changes from baseline after surgery. | Day 0, On Day1, and on Day 2 after surgery.
  Measurement of heart rate in Beat per minutes changes from baseline after surgery. On Day 0 after surgery, on Day1, and on Day2 after surgery.
Assessment of respiratory rate changes from baseline. | Day 0, On Day1, and on Day 2 after surgery.
  Measurement of respiratory rate in breath per minutes changes from baseline. On Day 0 after surgery, on Day1, and on Day2 after surgery.
Assessment of Oxygen saturation changes from baseline. | Day 0 after surgery, on Day1, and on Day2 after surgery.
  Measurement of oxygen saturation percentage changes from baseline. On Day 0 after surgery, on Day1, and on Day2 after surgery.
Noninvasive blood pressure changes from baseline after surgery. | Day 0 after surgery, on Day1, and on Day2 after surgery.
  Noninvasive Measurement of blood pressure after surgery in Milliliter of mercury changes from baseline. Measurement of Systolic and diastolic blood pressure changes on Day 0 after surgery, on Day1, and on Day2 after surgery.

SECONDARY OUTCOMES:
Post operative Pain score | On Day 0, On Day1, and on Day 2.
  Pain scale used are "Visual analogue score' for pain assessment at rest, and "visual analogue score' for pain assessment with movement. Pain scale scores (assessment during movement and during rest), are from 0 to 10. Pain score of 0 means no pain, which indicate that the 'Quadratus lumborum block is very effective (desired outcome). Pain score of 10 means worst imaginable pain, which indicate that the block is not effective (Undesired outcome).
Measurement of Time to mobilization in hours after surgery. | From 1st hour up to 48th hour after surgery.
  Recording of the time when the patient is able to stand on her legs and move out of the bed alone after the surgery. Time to mobilization in hours up to 48th hour after surgery. Early mobilization indicates successful block of pain after surgery without affecting lumber plexus nerves (desired outcome).
  Delayed mobilization indicates block extending to lumber plexus nerves (Undesired outcome).
Assessment of Nausea and Vomiting postoperative. | From 1st hour up to 48th hour after surgery.
  "Nausea scale", the Nausea scale score is from 0 to 3, when score of: 0 indicate No Nausea, score of 1 indicate mild nausea without vomiting, score of 2 indicate moderate nausea without vomiting, and score of 3 indicate severe nausea with vomiting (Undesired outcome).
  Assessment at hours 1st, 2nd, 4th, 8th, 12th, 24th, and at 48th hour after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Danat Al Emarat hospital, Abu Dhabi, United Arab Emirates

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT05643846/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT05643846/ICF_001.pdf